CLINICAL TRIAL: NCT04676620
Title: Comparison of Anterior Corneal Optical Aberration Induced by Conductive Keratoplasty and Hyperopic Laser in Situ Keratomileusis
Brief Title: Comparison of Anterior Corneal Optical Aberration Induced by CK and Hyperopic LASIK
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Wang Hongxia (Other)
Collaborators: Tianjin Eye Hospital (Other)
Responsible Party: Sponsor-Investigator, Wang Hongxia, Shanghai Guanghua Hospital of Integrated Traditional Chinese and Western Medicine, Shanghai Guanghua Hospital of Integrated Traditional Chinese and Western Medicine
Organization: Shanghai Guanghua Hospital of Integrated Traditional Chinese and Western Medicine (Other)
Other Study IDs: 2020-K-107
Record Dates: First submitted 2020-12-15; First posted 2020-12-21 (Actual); Last update posted 2020-12-21 (Actual); Status verified 2020-12

CONDITIONS: Refractive Error
Keywords: conductive keratoplasty; corneal optical aberrations; hyperopic corrections; LASIK
MeSH Terms: conditions — Refractive Errors

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- CK surgery: Conductive keratoplasty (CK) had shown to be a safe and effective procedure for the treatment of low to moderate hypeopia. It had been approved by the U.S. Food and Drug Administration (FDA) to treat presbyope in early 2004. CK appeals to both surgeons and patients as it avoids the need for flap creation, the use of high intraocular pressure (IOP), or tissue ablation.
  Interventions: Procedure: CK surgery
- LASIK surgery: LASIK surgery is femtosecond laser assisted conventional refractive surgery and has also been proved to offer many advantages in terms of visual acuity, corneal sensitivity, and corneal biomechanics compared with traditional refractive surgeries.
  Interventions: Procedure: CK surgery

INTERVENTIONS:
Procedure: CK surgery — CK and LASIK are both effective methods for the correction of hypeopia. They have been proved to offer many advantages in terms of visual acuity, corneal sensitivity, and corneal biomechanics compared with traditional refractive surgeries.

SUMMARY:
Conductive keratoplasty (CK) had shown to be a safe and effective procedure for the treatment of low to moderate hypeopia. It had been approved by the U.S. Food and Drug Administration (FDA) to treat presbyope in early 2004. CK appeals to both surgeons and patients as it avoids the need for flap creation, the use of high intraocular pressure (IOP), or tissue ablation. It utilizes "blended vision" rather than the true monovision used with laser in situ keratomileusis (LASIK), which patients tolerate more readily. There is very little reported research about the induction of wavefront aberration by CK. The symptomatology of high order aberrations (HOA) and the way individual Zernike functions were correlated with visual acuity, contrast sensitivity, visual symptoms. This study measured the HOA created by surgically induced myopic shift via CK and LASIK in an effort to better understand the phenomena of regression, multifocality, pseudo-accommodation and monovision.

DETAILED DESCRIPTION:
To investigate anterior corneal optical higher order aberration (HOA) induced by conductive keratoplasty (CK) and laser in situ keratomileusis (LASIK). 69 eyes with hyperopia or presbyopia were enrolled. 47 eyes of 47 patients underwent CK procedure, 22 eyes underwent LASIK. Data were acquired preoperatively, and at 3 and 6 months postoperatively. The total Root Mean Square (RMS) of the HOA as well as the individual Zernike polynomials of coma, trefoil, and spherical aberration were analyzed. In CK group, the high order RMS showed significant elevation at 3 months, but it returned to near preoperative levels at 6 months postoperatively. Trefoil (Z33) is the exclusive Zenike pattern to increase significantly following CK, peaking at 3 months and then decreasing back to near preoperative level at 6 months after CK. In the hyperopic LASIK group, coma increased to a peak at 3 month postoperatively, and persisted at sixth month after LASIK. Spherical aberration decreased significantly at 3 months and persisted till the sixth postoperative month. There was significant correlation between ΔSE and Δspherical aberration showed in both groups. The HOA and main Zernike polynomials pattern and their natural changes induced by CK is significantly different from that induced by LASIK in the hyperopic corrected treatment. The amount of achieved hyperopic corrections induced by CK or LASIK is not correlated to the change of HOA patterns such as coma and trefoil, but it is correlated to the change of spherical aberration.

ELIGIBILITY:
Inclusion Criteria:

* age of over 40 years old (yrs)
* stable refraction
* planned to induce a myopic shift

Exclusion Criteria:

* age of less than 40 years old (yrs)
* significant systemic illnesses
* congenital myopia,
* media opacity uveitis
* glaucoma
* intraocular surgery refractive surgery
* neurologic diseases
* retinal disease

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: In this consecutive case series, 69 eyes of 57 patients (30 female and 27 male) with hyperopia or presbyopia were enrolled. Inclusion criteria included age of over 40 years old (yrs), stable refraction, and patients who were planned to induce a myopic shift ranging of -1.00 diopters (D) to -2.50D. Mean patient age was 52.9±5.7 yrs (range from 42 to 68 yrs). The ophthalmic examination for each patient included uncorrected visual acuity (UCVA), best spectacle-corrected visual acuity (BSCVA) (Snellen chart), near vision (Jaeger chart), manifest and cycloplegic refraction, videokeratography, central and peripheral corneal ultrasound pachymetry (thickness), slit-lamp microscopy, dilated fundus examinations, IOP.
Sampling Method: Non-Probability Sample
Enrollment: 69 (Estimated)
Dates: Start 2020-12 (Estimated); Primary Completion 2021-12 (Estimated); Study Completion 2021-12 (Estimated)

PRIMARY OUTCOMES:
uncorrected visual acuity | change from baseline with EDTRS chart at 6 months
  uncorrected visual acuity change from baseline at 6 months
best spectacle-corrected visual acuity | change from baseline with EDTRS chart at 6 months
  best spectacle-corrected visual acuity change from baseline with EDTRS chart at 6 months

SECONDARY OUTCOMES:
near vision | change from baseline with EDTRS chart at 6 months
  near vision change from baseline with EDTRS chart at 6 months
central and peripheral corneal ultrasound pachymetry | change from baseline with EDTRS chart at 6 months
  central and peripheral corneal ultrasound pachymetry change from baseline with EDTRS chart at 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Hongxia Wang, director, Study Director — Shanghai Guanghua integrated traditional Chinese and Western Medicine Hospital
Locations (1):
- Shanghai Guanghua Integrated Traditional Chinese and Western Medicine Hospital, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Du TT, Fan VC, Asbell PA. Conductive keratoplasty. Curr Opin Ophthalmol. 2007 Jul;18(4):334-7. doi: 10.1097/ICU.0b013e3281df2cf0. PMID 17568211
- [Result] Lin DY, Manche EE. Two-year results of conductive keratoplasty for the correction of low to moderate hyperopia. J Cataract Refract Surg. 2003 Dec;29(12):2339-50. doi: 10.1016/j.jcrs.2003.09.022. PMID 14709295
- [Result] Pallikaris lG, Naoumidi TL, Panagopoulou SI, Alegakis AK, Astyrakakis NI. Conductive keratoplasty for low to moderate hyperopia: 1-year results. J Refract Surg. 2003 Sep-Oct;19(5):496-506. doi: 10.3928/1081-597X-20030901-04. PMID 14518738